CLINICAL TRIAL: NCT05433285
Title: Immunogenicity & Safety of SARS-CoV-2 Protein Subunit Recombinant Vaccine (Bio Farma) Adjuvanted With Alum+CpG 1018 Compared to Registered Covid-19 Vaccine (Covovax - Protein Subunit Vaccine) in Healthy Populations Aged 18 Years and Above in Indonesia (Phase III)
Brief Title: Immuno-bridging Study of COVID-19 Protein Subunit Recombinant Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Faculty of Medicine Universitas Diponegoro (Unknown); Faculty of Medicine Universitas Andalas (Unknown); Faculty of Medicine Universitas Hassanudin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CoV2-IB-0322
Record Dates: First submitted 2022-06-23; First posted 2022-06-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; healthy population; naive participants
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Vaccine candidate and active comparator are masking, lot number is masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Protein Subunit Recombinant Vaccine (Experimental): 2 doses of COVID-19 Protein Subunit Recombinant Vaccine administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: COVID-19 Protein Subunit Recombinant Vaccine
- Active Comparator (Active Comparator): 2 doses of Covovax® - recombinant spike protein Nanoparticle Vaccine, administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: Active Comparator

INTERVENTIONS:
Biological: COVID-19 Protein Subunit Recombinant Vaccine — SARS-CoV-2 RBD subunit recombinant protein, manufactured by PT. Bio Farma
  Arms: COVID-19 Protein Subunit Recombinant Vaccine
Biological: Active Comparator — Covovax® COVID-19 vaccine is a protein-based vaccine candidate engineered from the genetic sequence of the first strain of the SARS-CoV-2 betacoronavirus
  Arms: Active Comparator

SUMMARY:
Observer-blind, randomized, active-controlled prospective intervention study

DETAILED DESCRIPTION:
This trial is randomized, prospective intervention study. A total of 4,050 subjects (COVID-19 vaccine naive) who are willing to participate in the study by signing the consent form, will be involved in this trial. The subjects will be divided into three study subsets, namely Main Study I, Main Study II, and Exploratory Study: Main Study I for immunogenicity and safety evaluation, Main Study II for safety evaluation, and Exploratory Study for cellular immunity evaluation, with trial design as follow :

* Main Study I, Exploratory Study subset: Observer-blind, randomized, active-controlled prospective intervention study
* Main Study II: Open-label, randomized study to evaluate safety I

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects aged 18 years and above.
2. Subjects have been informed properly regarding the study and signed the informed consent form.
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. History of vaccination with any COVID-19 vaccine.
3. History of COVID-19 within 1 month (for mild-moderate disease) or 3 months (for severe disease) prior to enrollment.
4. Evolving mild, moderate, or severe illness, especially infectious disease, or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. Women who are pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
6. History of uncontrolled asthma, allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
7. History of blood disorders contraindicating intramuscular injection.
8. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc.) which according to the investigator might interfere with the assessment of the trial objectives.
9. History of confirmed or suspected immunosuppressive or immunodeficient state or in the previous 4 weeks received a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, or long-term corticosteroid therapy (> 2 weeks)).
10. History of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
11. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
12. Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4050 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the candidate vaccine | 14 days after the last dose
  Geometric Mean Titers (GMT) of neutralizing antibody
Seroconversion rate of the candidate vaccine | 14 days after the last dose
  Seroconversion rate of neutralizing antibody

SECONDARY OUTCOMES:
Safety of the candidate vaccine | 28 days after each dose
  percentage of subjects with solicited and unsolicited Adverse Events (AE)
Serious Adverse Event (SAE) of the vaccine | 12 months after the last dose
  percentage of subjects with at least 1 SAE
Persistence neutralizing antibody of vaccine candidate | 28 days, 3 months, 6 months and 12 months after the last dose
  GMT of neutralization antibody
Persistence Immunoglobulin G (IgG) antibody of vaccine candidate | 14 days, 28 days, 3 months, 6 months and 12 months after the last dose
  GMT of IgG antibody (RBD)

OTHER OUTCOMES:
Cellular immunity of candidate vaccine | 14 days, 6 months and 12 months after two-dose primary series.
  Positive rate of specific T-cell response

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Soedjatmiko SpA(K), MSi, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (4):
- Indonesia (4):
  - Faculty of Medicine Diponegoro University, Semarang, Central Java
  - Fakultas Kedokteran Universitas Indonesia, Jakarta, Greater Jakarta
  - Faculty of Medicine Universitas Hassanudin, Makassar, South Sulawesi
  - Faculty of Medicine Universitas Andalas, Padang, West Sumatera

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nurdin A, Movieta Nency Y, Maddeppungeng M, Sekartini R, Mulia Sari R, Surachman F, Fitry Yani F, Raveinal, Anggrainy F, Hafiz A, Linosefa, Machmud R, Awaliyah Deza P, Rujiana V, Bella Rahimi M, Farhanah N, Gundi Pramudo S, Hapsari R, Tri Anantyo D, Mulyono, Mahati E, Maharani N, Darma S, Husni Esa Darussalam A, Shakinah S, Nasrum Massi M, Soedjatmiko. Immunogenicity and safety of SARS-CoV-2 recombinant protein subunit vaccine (IndoVac) adjuvanted with alum and CpG 1018 in Indonesian adults: A phase 3, randomized, active-controlled, multicenter trial. Vaccine. 2024 Apr 30;42(12):3009-3017. doi: 10.1016/j.vaccine.2024.03.077. Epub 2024 Apr 4. PMID 38575433